CLINICAL TRIAL: NCT05891522
Title: Pilot Study of the Use of a Portable Cranial Scanner in Intensive Care for Cerebro-injured Patients
Acronym: ESPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC18_8960_ESPER; 2018-A02723-52 (Other: N°ID-RCB)
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Craniocerebral Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- portable scanner (Experimental)
  Interventions: Procedure: portable scanner
- fixed scanner (Active Comparator)
  Interventions: Procedure: fixed scanner

INTERVENTIONS:
Procedure: portable scanner — performing a portable cranial scanner on cerebro-injured intensive care patients
  Arms: portable scanner
Procedure: fixed scanner — performing a conventional fixed cranial scanner on cerebro-injured intensive care patients
  Arms: fixed scanner

SUMMARY:
Cerebral scans are a key examination in the management of serious brain-injured patients in intensive care, and are often repeated in the initial phase. This is a critical clinical period for these fragile patients, who are likely to develop episodes of intracranial hypertension (ICHT), the duration of which is correlated with a poor prognosis. These patients are therefore exposed to the complications of intra-hospital transport (IHT) (HTIC, hypoxaemia, arterial hypotension, disconnection of the respirator, respiratory asynchronies), which can worsen their vital and neurological prognosis. The incidence of adverse events linked to HIT has been estimated at up to 79.8%, including episodes of HTIC, worsening the prognosis and increasing the length of hospitalisation. In addition, patient safety during HIT requires the mobilisation of a doctor, a nurse and a care assistant, an organisation that implies a reduction in the care team's time with the other intensive care patients in their care. In this context, the portable cranial scanner, with imaging quality similar to that of conventional scanners, is already in routine use in the United States, the United Kingdom and Germany. This tool could reduce examination times, thereby reducing the risk of adverse events for the patient, in particular episodes of HTIC, and optimising the mobilisation of intensive care professionals. Studies suggest that the use of portable cranial scanners significantly reduces the duration of the examination (total duration including transport time) (50 minutes for conventional scanners versus 20 minutes for portable scanners), without altering the cerebral perfusion pressure or intracranial pressure of intensive care patients.

In addition, the use of portable scanners could generate savings for hospitals. In fact, in American and British teams where the use of portable scanners is widespread, several studies have shown that the time spent by radiology staff is reduced and the number of intensive care professionals mobilised is reduced compared with the use of conventional scanners. In addition, freeing up conventional scanner slots could lead to an increase in conventional scanner activity. For example, in a neurovascular emergency department environment at Massachusetts General Hospital, USA, the introduction of a mobile scanner reduced access time to the examination by 58% (39 minutes ±5.1 vs. 17 ±2.7 for conventional scanning), which also suggests faster implementation of emergency treatments such as the intravenous thrombolysis evaluated in this study. Finally, an American study carried out in 2008 estimated the financial gain generated by the use of a portable scanner versus a conventional scanner at more than 2 million dollars over 5 years and a complete return on investment of 7 months, from a hospital point of view.

To date, no French intensive care unit is using such a tool, even though the benefits appear to be real in terms of reducing the number of episodes of hypertensive haemorrhage and the prognostic impact this may have. The main aim of our pilot study is to assess the feasibility of using a portable brain scanner in cerebro-injured patients in intensive care by comparing the time taken to perform the portable examination with that of a conventional scanner. The investigators will also evaluate the existence and duration of HTIC episodes and the occurrence of any adverse events compared with a strategy based on a conventional fixed scanner.

ELIGIBILITY:
Inclusion Criteria:

* admitted to intensive care for moderate or severe head trauma or severe meningeal haemorrhage (Glasgow score < or = 12);
* need for a brain scan;

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Time taken to perform a cranial scan | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Launey, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France